CLINICAL TRIAL: NCT00656019
Title: Development of Vitamin D as a Therapy for Breast Cancer - Phase 2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Melinda Telli, Assistant Professor, Stanford University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-12226; 98671 (Other: Stanford University Alternate IRB Approval Number); BRSNSTU0026 (Other: OnCore Number)
Record Dates: First submitted 2008-04-04; First posted 2008-04-10 (Estimated); Results first posted 2017-12-02 (Actual); Last update posted 2017-12-02 (Actual); Status verified 2017-10

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Vitamin D; calcipotriene

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Normal Vitamin D Levels (No Intervention): No additional Vitamin D administered
- Low-normal Vitamin D Levels (Experimental): 2000 IU dose of Vitamin D per day administered orally
  Interventions: Drug: Vitamin D
- Low Vitamin D Levels (Experimental): 4000 IU dose of Vitamin D per day administered orally
  Interventions: Drug: Vitamin D
- Very-low Vitamin D Levels (Experimental): 6000 IU dose of Vitamin D per day administered orally
  Interventions: Drug: Vitamin D

INTERVENTIONS:
Drug: Vitamin D — 0, 2000, 4000, and 6000 IU per day orally
  Other Names: Calcipotriene
  Arms: Low Vitamin D Levels; Low-normal Vitamin D Levels; Very-low Vitamin D Levels

SUMMARY:
This study will assess whether levels of vitamin D impact the characteristics of a woman's breast cancer at diagnosis, and whether a short course of vitamin D in women with low levels of vitamin D changes the gene expression of their breast cancers.

DETAILED DESCRIPTION:
Patients undergoing core needle biopsy of breast abnormalities suspicious for breast cancer will be identified and enrolled in study. As well as those who have had a core needle biopsy demonstrating breast cancer, but who have not yet undergone local surgical treatment, chemotherapy, or hormonal therapy are also eligible. patients with breast cancer on core biopsy will be eligible.

Participants will be assigned to treatment (0, 2000, 4000, 6000 IU/day vitamin D by mouth) based solely on their serum vitamin D levels (Normal: >40 ng/mL; Low-normal: 31-40 ng/mL; Low: 20-30 ng/mL; Very-low: <20 ng/mL). Prior to definitive breast cancer surgery, vitamin D level, parathyroid level, and calcium will be reassessed. Samples of the patients original core biopsy and pathology specimen from their definitive surgical therapy will undergo gene expression profiling.

The ultimate plan is to correlate baseline vitamin D levels with classic prognostic and predictive markers to see if breast cancer biology is impacted by baseline vitamin D level and by vitamin D supplementation and to see if vitamin D supplementation results in gene expression changes similar to those of the vitamin D sufficient group.

ELIGIBILITY:
INCLUSION CRITERIA:

* Undergoing core needle biopsy for a breast abnormality suspicious for breast cancer.
* Has undergone a core needle biopsy demonstrating breast cancer and has not yet had any further therapy, provided the core needle biopsy is available for analysis.
* No prior therapy for breast cancer within the past 5 years.
* 18 years of age or older.
* Ability to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

* History of parathyroid disease, hypercalcemia, or kidney stones.
* Supplemental vitamin D other than from a standard multiple vitamin or from standard formulations of calcium and vitamin D (eg, calcium citrate with vitamin D) within the prior 6 months.
* History of renal failure requiring dialysis or kidney transplantation.
* Pregnant or nursing
* Receiving supplemental calcium > 1200 mg calcium per day during study.
* Initial treatment of breast cancer will not be with breast-conserving surgery or mastectomy.
* Locally-advanced breast cancer
* Plans for neoadjuvant chemotherapy, hormonal therapy, or other systemic therapy
* Plans for preoperative radiation therapy
* Plans for breast cancer surgery, and does not allow for at least 10 days of vitamin D intervention.
* Any condition potentially interfering with subjects ability to comply with taking study medication.
* Any medical condition that would potentially interfere with vitamin D absorption, such as celiac sprue, ulcerative colitis.
* Current participation in another research study that would increase risk to subject, in the opinion of the investigators

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2008-04; Primary Completion 2010-08 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melinda Telli, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Normal Vitamin D Levels | Low-normal Vitamin D Levels | Low Vitamin D Levels | Very-low Vitamin D Levels
Started | 29 | 19 | 11 | 4
Completed | 15 | 18 | 11 | 4
Not Completed | 14 | 1 | 0 | 0
Not completed — Not Eligible | 10 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0 | 0
Not completed — Lost to Follow-up | 2 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- No Intervention (No Vitamin D); 2000 UI Vitamin D; 4000 UI Vitamin D; 6000 UI Vitamin D: Patients with breast cancer detected by biopsy
- Total: Total of all reporting groups
Arm/Group | No Intervention (No Vitamin D) | 2000 UI Vitamin D | 4000 UI Vitamin D | 6000 UI Vitamin D | Total
Number analyzed (Participants) | 15 | 18 | 11 | 4 | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 5 | 11 | 9 | 3 | 28
  >=65 years | 10 | 7 | 2 | 1 | 20
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 18 | 11 | 4 | 48
  Male | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 1 | 1 | 4
  Not Hispanic or Latino | 14 | 17 | 8 | 2 | 41
  Unknown or Not Reported | 0 | 0 | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 3 | 2 | 1 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 1 | 1
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 13 | 15 | 7 | 2 | 37
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 2 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Correlation of Vitamin D Levels, Prognostic Factors, and Gene Expression Profile in Patients With Breast Cancer
Description: Vitamin D levels in serum were correlated to classic prognostic and predictive factors for breast cancer, and the gene expression profile of breast core biopsy specimens. The outcome is reported as the proportion of subjects with a discernible pattern for expression of the set of 40 evaluated genes
Time Frame: 10 days to 4 weeks post diagnosis.
Measure: Number; unit: percentage of participants
Arm/Group | Normal Vitamin D Levels | Low-normal Vitamin D Levels | Low Vitamin D Levels | Very-low Vitamin D Levels
Number analyzed (Participants) | 15 | 18 | 11 | 4
percentage of participants | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 3 Years
Groups:
- Vitamin D Normal: No Additional Vitamin D will be given (these patients have normal Vitamin D levels).
- Vitamin D Low-normal: 2000 IU dose of vitamin D per day (these patients have slightly low vitamin D levels).
  Vitamin D: 2000 IU per day orally
- Vitamin D Low: 4000 IU dose of vitamin D per day (these patients have low vitamin D levels).
  Vitamin D: 4000 IU per day orally
- Vitamin D Very Low: 6000 IU dose of vitamin D per day (these patients have very low vitamin D levels).
  Vitamin D: 6000 IU per day orally
Arm/Group | Vitamin D Normal | Vitamin D Low-normal | Vitamin D Low | Vitamin D Very Low
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/19 | 0/11 | 0/4
Other Adverse Events (participants affected / at risk) | 0/29 | 0/19 | 0/11 | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes